CLINICAL TRIAL: NCT06432101
Title: Clinical Efficacy of Acupuncture Combined With Hydroxychloroquine Sulfate Tablets in Improving Oral and Ocular Dryness in Primary Sjögren's Syndrome
Brief Title: Acupuncture Combined With Hydroxychloroquine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senyue Zhang (Other)
Responsible Party: Sponsor-Investigator, Senyue Zhang, Principal Investigator, Heilongjiang University of Chinese Medicine
Organization: Heilongjiang University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 595661170@qq.com
Record Dates: First submitted 2024-05-10; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Primary Sjögren's Syndrome
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture combined with hydroxychloroquine sulfate tablets (Active Comparator): Acupuncture combined with oral hydroxychloroquine sulfate tablets
  Interventions: Other: Acupuncture combined with oral hydroxychloroquine sulfate tablets
- oral hydroxychloroquine sulfate tablets (No Intervention): Oral hydroxychloroquine sulfate tablets (Shanghai Shangyao Sino-Western Pharmaceutical Co., LTD., Fenle, Sinopyma approval number H19990263, 0.1g x 14 tablets) were treated with 0.2g each time, twice a day, 4 weeks for 1 course of treatment, a total of 2 courses of treatment.

INTERVENTIONS:
Other: Acupuncture combined with oral hydroxychloroquine sulfate tablets — Acupuncture combined with oral hydroxychloroquine sulfate tablets
  Arms: acupuncture combined with hydroxychloroquine sulfate tablets

SUMMARY:
To observe the clinical efficacy of acupuncture combined with hydroxychloroquine sulfate tablets on the symptoms of dry mouth and dry eyes in primary Sjögren's syndrome.

DETAILED DESCRIPTION:
Methods: Seventy-two patients with primary Sjögren's syndrome who met the inclusion criteria were randomly divided into the experimental group (36 patients, 3 patients who fell out) and the control group (36 patients, 4 patients who fell out). The control group was treated with oral hydroxychloroquine sulfate tablets alone, 0.2g each time, taken twice a day, 4 weeks for 1 course of treatment, a total of 2 courses of treatment, and the experimental group was treated with acupuncture treatment on the basis of the control group, acupuncture once a day, acupuncture for 5 days and 2 days of rest, 4 weeks for 1 course of treatment, a total of 2 courses of treatment. The changes in the outcome indicators of the two groups before and after treatment were observed, and the main outcome indicators included salivary flow rate (SFR) and Schirmer test. Secondary outcomes included the European League Against Rheumatism (EULAR) Sjögren's Syndrome Patient-Reported Index (ESSPRI), the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI), and laboratory measures (ESR, CRP, IgG).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary Sjögren's syndrome
* Must be able to receive acupuncture treatment and swallow tablets

Exclusion Criteria:

* Patients with malignant tumors or severe organ function impairment
* Patients who are lactating or pregnant.
* Persons who are participating in clinical trials of other drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Salivary flow rate (Sauf) | 8 weeks
  Used to evaluate the salivary flow rate of pSS patients before and after treatment. Before the start of the experiment, the patient gargled with water to keep the mouth clean and free of irritation. Saliva collected at the bottom of the mouth and spit it into the measuring cup every 1min. After collecting it for 10min, the value was recorded. The less the saliva flow rate within 10 minutes, the worse the symptoms, and less than 1ml is abnormal.
Schirmer test | 8 weeks
  Used to evaluate the degree of tear secretion in pSS patients before and after treatment. The 5mm×35mm filter paper was folded at a right Angle at 5mm from one end, and the end was placed in the conjunctival sac at 1/3 of the outer eyelid of the patient. The eyes were closed and the clamp was held for 5min, and the wet length of the filter paper was measured, and the filter paper was positive if it was less than 5mm/5min. The less tears are secreted within five minutes, the more severe the symptoms.

SECONDARY OUTCOMES:
Sjögren's syndrome patient-reported index (ESSPRI) | 8 weeks
  Used to assess the degree of dryness, pain, and fatigue in pSS patients, it is an evaluation of disease activity based on patients' subjective feelings. On a scale of 0 to 10 from mild to severe, the final ESSPRI score is the average score of dryness, pain and fatigue. Scores <5 were classified as acceptable symptom status and >5 as unsatisfactory symptom status.
EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) score | 8 weeks
  used to evaluate disease activity in patients with pSS, ESSDAI is an evaluation of disease activity based on objective facts. The score weight includes 12 dimensions, including systemic symptoms, lymph node disease, glandular disease, joint disease, skin disease, peripheral neuropathy, central neuropathy, lung disease, kidney disease, muscle disease, hematological diseases and serological changes. The total score of ESSDAI is equal to the sum of the score of the severity of each system × the product of the weight of the system. A scale of <5 was classified as low disease activity, 5 to 13 as moderate disease activity, and >14 as high disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Senyue Zhang, Principal Investigator — Heilongjiang University of Chinese Medicine
Locations (1):
- Senyue Zhang, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No